CLINICAL TRIAL: NCT05370040
Title: THEMBA II T-CELL Vaccine: A Phase 1/2 Study of the Safety, Reactogenicity, and Immunogenicity of Vaccination With saRNA COVID-19 Vaccines
Brief Title: THEMBA II T-Cell Vaccine: Vaccination With saRNA COVID-19 Vaccines
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinued prior to enroll in Phase 2
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: COVID-4.015
Record Dates: First submitted 2022-05-09; First posted 2022-05-11 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Emergency Use Authorization

STUDY DESIGN:
Intervention Model Description: Open label 6 Cohort Phase 1 Study leading to Randomized 4 Cohort Phase 2 Study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Phase 1 Cohort 1A (Experimental): AAHI-SC2 on Day 1 at dosage 25 μg IM
  Interventions: Biological: AAHI-SC2 Vaccine
- Phase 1 Cohort 1B (Experimental): AAHI-SC2 on Day 1 at dosage 50 μg IM
  Interventions: Biological: AAHI-SC2 Vaccine
- Phase 1 Cohort 1C (Experimental): AAHI-SC2 on Day 1 at dosage 70 μg IM
  Interventions: Biological: AAHI-SC2 Vaccine
- Phase 1 Cohort 2A (Experimental): AAHI-SC3 on Day 1 at dosage 25 μg IM
  Interventions: Biological: AAHI-SC3 Vaccine
- Phase 1 Cohort 2B (Experimental): AAHI-SC3 on Day 1 at dosage 50 μg IM
  Interventions: Biological: AAHI-SC3 Vaccine
- Phase 1 Cohort 2C (Experimental): AAHI-SC3 on Day 1 at dosage 85 μg IM
  Interventions: Biological: AAHI-SC3 Vaccine
- Phase 2 Control arm (Placebo Comparator): EUA or approved vaccine on Day 1
  Interventions: Biological: EUA or approved vaccine
- Phase 2 Experimental arm 1 (Experimental): AAHI-SC2 on Day 1 Dose TBD as determined in phase 1 study
  Interventions: Biological: AAHI-SC2 Vaccine
- Phase 2 Experimental arm 2 (Experimental): AAHI-SC3 on Day 1 Dose TBD as determined in phase 1 study
  Interventions: Biological: AAHI-SC3 Vaccine
- Phase 2 Experimental arm 3 (Experimental): AAHI-SC3 on Day 1 and 29 Dose TBD as determined in phase 1 study
  Interventions: Biological: AAHI-SC3 Vaccine

INTERVENTIONS:
Biological: AAHI-SC2 Vaccine — AAHI -SC2 self-amplifying RNA (saRNA) against SARS-CoV-2 Spike protein delivered by nanostructured lipid carrier (NLC) Vaccine
  Arms: Phase 1 Cohort 1A; Phase 1 Cohort 1B; Phase 1 Cohort 1C; Phase 2 Experimental arm 1
Biological: AAHI-SC3 Vaccine — AAHI-SC3 self-amplifying RNA (saRNA) against SARS-CoV-2 Spike and nucleocapsid protein delivered by nanostructured lipid carrier (NLC) Vaccine
  Arms: Phase 1 Cohort 2A; Phase 1 Cohort 2B; Phase 1 Cohort 2C; Phase 2 Experimental arm 2; Phase 2 Experimental arm 3
Biological: EUA or approved vaccine — Janssen or Pfizer vaccines (control arm)
  Arms: Phase 2 Control arm

SUMMARY:
This is a phase 1/2 open-label study assessing the safety, reactogenicity, and immunogenicity of saRNA COVID-19 boost vaccines in participants that have been previously vaccinated against or previously infected with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults ≥ 18 years of age at time of enrollment.
2. Vaccinated with an EUA or approved vaccine against COVID-19 ≥ 3 months prior to enrollment on study or infection with COVID-19 ≥ 3 months prior to enrollment on study.
3. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
4. Agrees to the collection of biospecimens (eg, nasopharyngeal [NP] swabs) and venous blood per protocol.
5. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
6. Temperature < 38°C.
7. Agreement to practice effective contraception for female participants of childbearing potential and non-sterile males. Female participants of childbearing potential must agree to use effective contraception while on study until at least 1 month after the last dose of vaccine. Non-sterile male participants must agree to use a condom while on study until at least 1 month after the last dose of vaccine. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm), intrauterine devices (IUDs), oral contraceptives, injectable contraceptives, patches, implants and abstinence.
8. HIV-positive participants must have been on anti-retroviral therapy for ≥ 4 weeks and have HIV-1 viral load < 1,000 copies/mL at the time of enrollment.

Exclusion Criteria:

1. Serious adverse reaction to any vaccine, any unrelated medication or any component of the investigational vaccine, including a history of anaphylaxis and symptoms of a severe allergic reaction and history of allergies in the past.
2. Confirmed current COVID-19, previous SARS-CoV-2 infection in the last < 3 months, or PCR positive for SARS-CoV-2 at screening.
3. Vaccinated with an EAU-approved vaccine against COVID-19 in the last < 3 months.
4. Pregnant or breastfeeding women.
5. Chronic lung disease (included COPD) as evidenced by one or more exacerbations requiring a course of steroids in the last year, or the requiring chronic low dose oral steroids to prevent exacerbations. Uncontrolled asthma, defined as requiring reliever inhaler (short-acting beta agonist or ipratromium bromide) more than twice a week is also excluded.
6. Bone marrow or organ transplant recipient
7. Extreme obesity (defined as BMI of 40 kg/m2 or higher).
8. Chronic kidney disease requiring dialysis.
9. History of liver disease.
10. Any disease associated with acute fever, or any infection.
11. Participants with acquired or hereditary immunodeficiencies other than well-controlled HIV are excluded from enrollment.
12. Current diagnosis of active tuberculosis.
13. History of hereditary, idiopathic or acquired angioedema.
14. No spleen or functional asplenia.
15. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, or immunomodulators. The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.
16. According to the judgement of the investigator any medical, psychiatric, psychological, social, occupational or other conditions that could affect the participants ability to sign informed consent, provide safety assessment data or comply with the requirements of the study protocol.
17. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wits Vida, Johannesburg, South Africa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 9 | 10 | 9 | 10
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (12.52) | 28.7 (7.53) | 32.6 (9.00) | 37.2 (7.10) | 32.7 (11.44) | 29.3 (7.48) | 32.7 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 5 | 6 | 10 | 45
  Male | 2 | 2 | 2 | 5 | 4 | 0 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 10 | 10 | 10 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 10 | 10 | 10 | 10 | 10 | 60
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Healthy adults vaccinated with an EUA or approved vaccine against COVID-19 ≥3 months prior to enroll [Count of Participants; unit: Participants] | 10 | 10 | 10 | 10 | 10 | 10 | 60

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Safety - Incidence of MAAEs Through 1 Week
Description: Incidence of medically-attended adverse events (MAAEs)
Time Frame: through 1 week post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 1 | 2 | 1 | 0 | 0 | 0

2. Primary Outcome: Phase 1 Safety - Incidence of MAAEs Through 30 Days
Description: Incidence of MAAEs
Time Frame: through 30 days post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 2 | 2 | 2 | 2 | 0 | 1

3. Primary Outcome: Phase 1 Safety - Incidence of MAAEs Through 6 Months
Description: Incidence of MAAEs
Time Frame: through 6 months post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 5 | 3 | 2 | 2 | 2 | 2

4. Primary Outcome: Phase 1 Safety - Incidence of Solicited Local Reactogenicity AEs
Description: Incidence and severity of solicited local reactogenicity AEs
Time Frame: through 1 week after each vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 9 | 9 | 9 | 8 | 9 | 9

5. Primary Outcome: Phase 1 Safety - Incidence of Solicited Systemic Reactogenicity AEs
Description: Incidence and severity of solicited systemic reactogenicity AEs
Time Frame: through 1 week after each vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 9 | 10 | 10 | 8 | 9 | 9

6. Primary Outcome: Phase 1 Safety - Incidence of Unsolicited AEs Through 1 Week
Description: Incidence and severity of unsolicited AEs
Time Frame: through 1 week post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 4 | 1 | 1 | 1 | 1 | 3

7. Primary Outcome: Phase 1 Safety - Incidence of Unsolicited AEs Through 30 Days
Description: Incidence and severity of unsolicited AEs
Time Frame: through 30 days post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 5 | 2 | 5 | 4 | 5 | 7

8. Primary Outcome: Phase 1 Safety - Incidence of SAEs Through 1 Week
Description: Incidence of serious adverse events (SAEs)
Time Frame: through 1 week post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Phase 1 Safety - Incidence of SAEs Through 30 Days
Description: Incidence of SAEs
Time Frame: through 30 days post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 1 | 0 | 0

10. Primary Outcome: Phase 1 Safety - Incidence of SAEs Through 6 Months
Description: Incidence of SAEs
Time Frame: through 6 months post final vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: For 30 days after the last dose, at each study visit, the Investigator was to inquire about the occurrence of AE/SAEs since the last visit or follow-up. From 30 days after the last dose to 6 months after the last dose, at each study visit, the Investigator was to inquire about the occurrence of SAEs since the last visit or follow-up. Events were to be followed for outcome information until resolution or stabilization.
Groups:
- Group 1: Cohort 1A; Group 1: Cohort 1B; Group 1: Cohort 1C; Group 1: Cohort 2A; Group 1: Cohort 2B; Group 1: Cohort 2C: Incidence of Solicited Local Reactogenicity Adverse Events Through 1 Week Post Final Vaccine Administration
- Group 2: Cohort 1A; Group 2: Cohort 1B; Group 2: Cohort 1C; Group 2: Cohort 2A; Group 2: Cohort 2B; Group 2: Cohort 2C: Incidence of Solicited Systemic Reactogenicity Adverse Events Through 1 Week Post Final Vaccine Administration
- Group 3: Cohort 1A; Group 3: Cohort 1B; Group 3: Cohort 1C; Group 3: Cohort 2A; Group 3: Cohort 2B; Group 3: Cohort 2C: Incidence of Unsolicited Adverse Events Through 30 Days Post Final Vaccine Administration
- Group 4: Cohort 1A; Group 4: Cohort 1B; Group 4: Cohort 1C; Group 4: Cohort 2A; Group 4: Cohort 2B; Group 4: Cohort 2C: Incidence of Medically Attended Adverse Events Through 6 Months Post Final Vaccine Administration
Arm/Group | Phase 1 Cohort 1A | Phase 1 Cohort 1B | Phase 1 Cohort 1C | Phase 1 Cohort 2A | Phase 1 Cohort 2B | Phase 1 Cohort 2C | Group 1: Cohort 1A | Group 1: Cohort 1B | Group 1: Cohort 1C | Group 1: Cohort 2A | Group 1: Cohort 2B | Group 1: Cohort 2C | Group 2: Cohort 1A | Group 2: Cohort 1B | Group 2: Cohort 1C | Group 2: Cohort 2A | Group 2: Cohort 2B | Group 2: Cohort 2C | Group 3: Cohort 1A | Group 3: Cohort 1B | Group 3: Cohort 1C | Group 3: Cohort 2A | Group 3: Cohort 2B | Group 3: Cohort 2C | Group 4: Cohort 1A | Group 4: Cohort 1B | Group 4: Cohort 1C | Group 4: Cohort 2A | Group 4: Cohort 2B | Group 4: Cohort 2C
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 1/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 9/10 | 9/10 | 9/10 | 8/10 | 9/10 | 9/10 | 9/10 | 10/10 | 10/10 | 8/10 | 9/10 | 9/10 | 5/10 | 2/10 | 5/10 | 4/10 | 5/10 | 7/10 | 5/10 | 3/10 | 2/10 | 2/10 | 2/10 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1A (N=10) | Phase 1 Cohort 1B (N=10) | Phase 1 Cohort 1C (N=10) | Phase 1 Cohort 2A (N=10) | Phase 1 Cohort 2B (N=10) | Phase 1 Cohort 2C (N=10) | Group 1: Cohort 1A (N=10) | Group 1: Cohort 1B (N=10) | Group 1: Cohort 1C (N=10) | Group 1: Cohort 2A (N=10) | Group 1: Cohort 2B (N=10) | Group 1: Cohort 2C (N=10) | Group 2: Cohort 1A (N=10) | Group 2: Cohort 1B (N=10) | Group 2: Cohort 1C (N=10) | Group 2: Cohort 2A (N=10) | Group 2: Cohort 2B (N=10) | Group 2: Cohort 2C (N=10) | Group 3: Cohort 1A (N=10) | Group 3: Cohort 1B (N=10) | Group 3: Cohort 1C (N=10) | Group 3: Cohort 2A (N=10) | Group 3: Cohort 2B (N=10) | Group 3: Cohort 2C (N=10) | Group 4: Cohort 1A (N=10) | Group 4: Cohort 1B (N=10) | Group 4: Cohort 1C (N=10) | Group 4: Cohort 2A (N=10) | Group 4: Cohort 2B (N=10) | Group 4: Cohort 2C (N=10)
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1A (N=10) | Phase 1 Cohort 1B (N=10) | Phase 1 Cohort 1C (N=10) | Phase 1 Cohort 2A (N=10) | Phase 1 Cohort 2B (N=10) | Phase 1 Cohort 2C (N=10) | Group 1: Cohort 1A (N=10) | Group 1: Cohort 1B (N=10) | Group 1: Cohort 1C (N=10) | Group 1: Cohort 2A (N=10) | Group 1: Cohort 2B (N=10) | Group 1: Cohort 2C (N=10) | Group 2: Cohort 1A (N=10) | Group 2: Cohort 1B (N=10) | Group 2: Cohort 1C (N=10) | Group 2: Cohort 2A (N=10) | Group 2: Cohort 2B (N=10) | Group 2: Cohort 2C (N=10) | Group 3: Cohort 1A (N=10) | Group 3: Cohort 1B (N=10) | Group 3: Cohort 1C (N=10) | Group 3: Cohort 2A (N=10) | Group 3: Cohort 2B (N=10) | Group 3: Cohort 2C (N=10) | Group 4: Cohort 1A (N=10) | Group 4: Cohort 1B (N=10) | Group 4: Cohort 1C (N=10) | Group 4: Cohort 2A (N=10) | Group 4: Cohort 2B (N=10) | Group 4: Cohort 2C (N=10)
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 9 | 8 | 7 | 9 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 5 | 3 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site hypoaesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 4 | 5 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 4 | 3 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5 | 5 | 2 | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 5 | 3 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 9 | 9 | 6 | 8 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 8 | 5 | 8 | 8 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 10 | 10 | 6 | 8 | 7 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 4 | 4 | 6 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 4 | 2 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0 | 4 | 3 | 3 | 1 | 1 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early. Only the safety data is provided.

Only one adverse event table per AE category was presented to reduce data entry redundancy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: part 1 (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT05370040/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: part 2 (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT05370040/Prot_SAP_002.pdf